CLINICAL TRIAL: NCT07052409
Title: Developing Interventions for Protecting HIV-Exposed Uninfected Infants Against Severe Infections
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Adriana Weinberg, Professor of Pediatrics, Medicine and Pathology, University of Colorado, Denver
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24-1383 COMIRB
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Gut Microbiome
Keywords: Gut microbiome; HIV-exposed uninfected infant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inkomasi (Active Comparator): Diet supplementation with pasteurized fermented milk
  Interventions: Dietary Supplement: Inkomazi
- Control (No Intervention): No intervention

INTERVENTIONS:
Dietary Supplement: Inkomazi — Pasteurized fermented milk
  Arms: Inkomasi

SUMMARY:
Research has shown that babies who are exposed to HIV, but are uninfected (negative HIV status), have a bigger risk of developing severe infections. There are naturally occurring organisms in the gut that may determine how the body protects itself against infections. These organisms may be different in babies who were exposed to the HIV virus in utero, compared to those who were not exposed. This study wants to see if the organisms in the gut of babies can be modified by supplementing the diet of the pregnant mother or of the baby at 6 months of age with Inkomasi (pasteurized fermented milk). The study will compare the type and amount of organisms in those who received supplementation and those who did not receive supplementation.

DETAILED DESCRIPTION:
1. The study will enroll 24 pregnant women with HIV at 36 weeks gestational age and randomize them 1:1 to receive 500 ml daily of pasteurized fermented milk (Inkomasi) or not. Changes in maternal gut microbiota from enrollment to 2-4 weeks postpartum will be compared between groups. The study will also compare the gut microbiome at infants born to mothers who received Inkomasi with those born to mothers who did not receive Inkomasi.
2. The study will enroll 24 HIV-exposed uninfected infants (HEU) at 24 weeks of age and randomize them 1:1 to receive ≥15 ml daily of pasteurized fermented milk (Inkomasi) or not. Changes in infant gut microbiota from enrollment to 4 weeks after enrollment will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with HIV HIV-exposed uninfected infants

Exclusion Criteria:

-

Ages: 6 Months to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Infant gut microbiome | from enrollment to 4-10 weeks after enrollment
  16s rRNA and metagenomic sequencing
Maternal gut microbiome | 4-10 weeks after initiation of the intervention
  Shotgun metagenomics and 16s rRNA

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Weinberg, MD, Principal Investigator — AMC UCD
Locations (1):
- Witwatersrand, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: Yes
NICHD database
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After study publication
Access Criteria: Demographic information will be deposited in the NICHD public database. Raw 16S rRNA gene sequences and shotgun metagenomic sequences, along with associated metadata, will be deposited in SRA following MIMARKS standard.
  External investigators will be able to access the data using standard search methods.